CLINICAL TRIAL: NCT03143621
Title: The Effect of Coffee Consumption on Return to Bowel Function After Small Bowel Resection
Brief Title: The Effect of Coffee After Resection of Small Bowel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Carmel Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Coffee Small Bowel
Record Dates: First submitted 2017-04-18; First posted 2017-05-08 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Postoperative Ileus
MeSH Terms: interventions — Coffee; Water

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group, controlled clinical trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will not be told what group they are assigned to, however, complete masking will be difficult to achieve. The patient's treatment assignment is part of the medical record.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coffee (Experimental): 100 cc's of coffee administered three times per day until return to bowel function has been established.
  Interventions: Dietary Supplement: Coffee
- Water (Placebo Comparator): 100 cc's of warm water administered three times per day until return to bowel function has been established.
  Interventions: Other: Water

INTERVENTIONS:
Dietary Supplement: Coffee — Brewed, caffeinated coffee, 100 cc's each dose
  Arms: Coffee
Other: Water — Tap water heated to same temperature as coffee
  Arms: Water

SUMMARY:
Post-operative ileus ("post-op ileus") is a condition which can occur after surgery. This means that the bowels stop working correctly and food and liquids will not pass through in the normal manner. Post-op ileus can be uncomfortable and require a longer hospital stay until the bowels begin to function correctly again. Currently there are no effective methods for preventing post-op ileus. Some studies suggest there is a benefit from drinking coffee following colon or gynecological cancer surgeries with very little risk. However, the effects of coffee following small bowel surgery have not been studied. This randomized, controlled trial will compare the outcomes of patients who receive coffee during their hospital stay after small bowel surgery to similar patients who receive warm water. About 60 patients will be in each group. The main outcomes are time until the nasogastric tube is removed and length of hospital stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing small bowel resection. Can be elective, urgent or emergent.

Exclusion Criteria:

* Patient with atrial fibrillation who is considered a non-coffee drinker (drinks coffee less than 3 days per week over the last 4 weeks)
* Patients undergoing colon resection without removal of any portion of small bowel.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Time to removal of nasogastric tube | From date of hospital admission up to date of hospital discharge (anticipated up to 2 weeks)
  Time at placement to Time at removal through study completion

SECONDARY OUTCOMES:
Time to return of bowel function | From date of hospital admission up to date of hospital discharge (anticipated up to 2 weeks)
  Time from end of surgery to Time of first flatus or bowel movement through study completion
Length of Stay | From date of hospital admission up to date of hospital discharge (anticipated up to 2 weeks)
  Time from end of surgery to Time discharge order written

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Aguila, MD, Principal Investigator — Mount Carmel Health System
Locations (1):
- Mount Carmel Health System, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual patient data at this time.